CLINICAL TRIAL: NCT06597409
Title: Respiratory Muscle Stretching as an Adjunct to Pulmonary Rehabilitation: Outcomes in Chest Expansion, Dyspnea, and Cough in Post-Tuberculosis Bronchiectasis
Brief Title: Respiratory Muscle Stretching for Improving Chest Expansion and Dyspnea in Post-Tuberculosis Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IKFR-202408.03
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Bronchiectasis Post-Tuberculosis Lung Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Active Comparator): Group A (Standard Pulmonary Rehabilitation)
  Interventions: Other: Standard PR
- Experimental (Experimental): Group B (Standard PR + RMS)
  Interventions: Other: Standard PR plus Respiratory Muscle Stretching (RMS)

INTERVENTIONS:
Other: Standard PR — (Aerobic exercise, PLB, ACBT, Education)
  Arms: Active Comparator
Other: Standard PR plus Respiratory Muscle Stretching (RMS) — Standard PR plus Respiratory Muscle Stretching (RMS)
  Arms: Experimental

SUMMARY:
This study intends to examine the effectiveness of adding RMS to a traditional program of pulmonary rehabilitation regarding chest expansion, dyspnea, and cough symptoms in bronchiectasis post-tuberculosis patients. Bronchiectasis, resulting from tuberculosis treatment, is characterized by restricted chest wall motility, chronic dyspnea, and an irritating cough, factors that severely impair these patients' quality of life. It is assumed that RMS improves the compliance of the chest wall, thereby enhancing respiratory mechanics and consequently reducing symptoms. The outcomes will be compared between two groups: one group with standard pulmonary rehabilitation and another group with additional RMS exercises.

DETAILED DESCRIPTION:
Bronchiectasis involves the irreversible dilation and damage of the bronchi, forming an important long-term sequela in patients who have completed treatment for lung tuberculosis. This condition leads to restricted chest expansion, severe shortness of breath, and chronic cough, causing considerable distress to the affected patients' quality of life. Pulmonary rehabilitation, through aerobic exercise and breathing techniques such as Pursed Lip Breathing (PLB) and the Active Cycle of Breathing Technique (ACBT), has shown benefits in managing these symptoms. The potential additional benefit of exercises involving accessory respiratory muscles to improve chest wall mobility, using Respiratory Muscle Stretching (RMS) exercises, has not been well-explored. This single-blind randomized controlled trial will compare the effects of standard pulmonary rehabilitation alone versus standard rehabilitation combined with RMS exercises in patients with bronchiectasis post-tuberculosis. Outcomes will focus on changes in chest expansion, dyspnea, cough symptoms, and lung function parameters such as FEV1, FVC, and FEV1/FVC ratio. The study will involve 48 participants who meet the inclusion criteria and will run for four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* History of lung TB treatment
* Clinical or radiological diagnosis of bronchiectasis
* mMRC Dyspnea Scale grade 1-3

Exclusion Criteria:

* Pneumothorax
* Pleural effusion
* COVID-19
* Lung malignancy
* Chronic obstructive pulmonary disease
* Neuromuscular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Chest Expansion | 4 weeks
  Measured in centimeters at three different levels of the rib cage (upper, middle, and lower chest). An expansion of more than and equal to 3 cm is considered normal chest, and less than 3 cm is considered abnormal chest expansion in all three levels.

SECONDARY OUTCOMES:
Dyspnea | 4 weeks
  Assessed using the modified Medical Research Council Dyspnea Scale (mMRC) The mMRC comprises the following four scales: 0, no breathlessness except on strenuous exercise; 1, shortness of breath when hurrying on the level or walking up a slight hill; 2, walks slower than people of same age on the level because of breathlessness or has to stop to catch breath when walking at their own pace on the level; 3, stops for breath after walking approximately 100 meters or after few minutes on the level; and 4, too breathless to leave the house, or breathless when dressing or undressing.
Cough Symptoms | 4 weeks
  Assessed using the modified Medical Research Council Dyspnea Scale (mMRC) The mMRC comprises the following four scales: 0, no breathlessness except on strenuous exercise; 1, shortness of breath when hurrying on the level or walking up a slight hill; 2, walks slower than people of same age on the level because of breathlessness or has to stop to catch breath when walking at their own pace on the level; 3, stops for breath after walking approximately 100 meters or after few minutes on the level; and 4, too breathless to leave the house, or breathless when dressing or undressing.
Forced Vital Capacity (FVC) | 4 weeks
  Lung function Forced Vital Capacity (FVC) is commonly assessed through spirometry and measured in liters (L) FVC: This measures the total volume of air that can be forcibly exhaled after a full inhalation.
  FVC values less than 80% of the predicted value are indicative of restrictive respiratory impairments, where the lungs cannot fully expand. FVC values equal to or greater than 80% are considered normal.
Forced Expiratory Volume in one second (FEV1) | 4 weeks
  Lung function Forced Expiratory Volume in one second (FEV1) is commonly assessed through spirometry and measured in liters (L) FEV1: This represents the air volume a person can forcefully exhale in the first second of a breath.
Ratio FEV1 and FVC | 4 weeks
  Lung function specifically the ratio of FEV1 and FVC (FEV1/FVC) is commonly assessed through spirometry and expressed as a percentage (%) FEV1/FVC: It is a key indicator of lung function. A normal FEV1/FVC ratio is typically greater than or equal to 70%. A ratio below this threshold suggests obstructive lung diseases, whereas a ratio above 70% but with reduced lung volumes may indicate restrictive lung diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Dian Marta Sari, MD., M.Sc., Ph.D, Principal Investigator — Faculty of Medicine Universitas Padjadjaran Bandung
Locations (1):
- Dr. M. Goenawan Partowidigdo Lung Hospital, Bogor, West Java, Indonesia